CLINICAL TRIAL: NCT03993821
Title: An Open Label Trial to Assess the Safety and Efficacy of Burosumab in a Single Patient With Cutaneous Skeletal Hypophosphatemia Syndrome (CSHS)
Brief Title: Burosumab for CSHS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laura Tosi (Other)
Collaborators: Children's National Research Institute (Other); Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Laura Tosi, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 11746
Record Dates: First submitted 2019-02-13; First posted 2019-06-21 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Cutaneous Skeletal Hypophosphatemia Syndrome (CSHS); Epidermal Nevus Syndrome
Keywords: CSHS; Cutaneous Skeletal Hypophosphatemia Syndrome; Epidermal Nevus Syndrome
MeSH Terms: conditions — Nevus, Sebaceous of Jadassohn | interventions — burosumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, 52-week study designed to assess the efficacy, safety and pharmacodynamics (PD) of burosumab in a single subject with cutaneous skeletal hypophosphatemia syndrome (CSHS). Burosumab (formerly KRN23) is a fully human immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that binds to and inhibits the activity of fibroblast growth factor 23 (FGF23), leading to an increase in serum phosphorus levels. It is hypothesized that burosumab may provide clinical benefit in this patient due to the common underlying feature in this patient and in patients with X-linked hypophosphatemia (in whom burosumab is FDA-approved) - abnormally elevated FGF23, in the context of low age-adjusted serum phosphorous levels. Patient will be seen at Screening, Baseline and every 2-4 wks, as described in "Schedule of Activities"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Burosumab (Experimental): Burosumab, which is FDA-approved for X-linked hypophosphatemic rickets, will be given monthly, for a total of 12 months and titrated to achieve a target fasting serum phosphorus level within normal range for age. The chosen starting dose of burosumab will be 0.3 mg/kg given SQ Q4W. The maximum dose allowed in this protocol is 2.0 mg/kg. Burosumab will be administered via subcutaneous (SC) route.
  Interventions: Drug: Burosumab

INTERVENTIONS:
Drug: Burosumab — Burosumab, the investigational product, is a recombinant human IgG1 monoclonal antibody targeting FGF23. It is supplied as a sterile, clear, colorless and preservative-free solution and is administered via subcutaneous injection.
  Other Names: Crysvita

SUMMARY:
Burosumab (also known as the drug, Crysvita®) is a fully human immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that binds to and inhibits the activity of fibroblast growth factor 23 (FGF23), leading to an increase in serum phosphorus levels. This drug is already approved for use in patients with X-linked hypophosphatemia (XLH), but not for Cutaneous Skeletal Hypophosphatemia Syndrome (CSHS). It is hypothesized that burosumab may provide clinical benefit to a patient with CSHS due to the common underlying feature in this patient and in patients with XLH - abnormally elevated FGF23 in the context of low age -adjusted serum phosphorous levels.

DETAILED DESCRIPTION:
There are multiple disorders (each with a unique underlying cause) that result in unusually high circulating levels of FGF23, which in turn result in renal phosphate wasting and reduced (or aberrantly normal in relationship to elevated FGF23) levels of 1,25-dihydroxy vitamin D (1,25[OH]2D). Across these disorders the clinical symptoms are similar and often include osteomalacia (and, in children, rickets), muscle weakness, fatigue, bone pain, and fractures. Burosumab has been FDA-approved for one of these disorders, X-linked hypophosphatemia (XLH). In single- and repeat-dose clinical studies in subjects with XLH, subcutaneous (SC) administration of burosumab consistently increased and sustained serum phosphorus levels and tubular reabsorption of phosphate (TRP) and improved radiologic rickets, without a major impact on urine calcium levels. Positive results were also observed in a nonclinical pharmacology model of XLH. It is hypothesized that burosumab may provide clinical benefit in this patient due to the common underlying feature in this patient and in patients with XLH - abnormally elevated FGF23 in the context of low age -adjusted serum phosphorous levels.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Patient has confirmed CSHS by physician diagnosis
2. Patient has confirmed FGF23 elevations in the context of a low fasting serum phosphorous < 2.5 mg/dL
3. Patient able to tolerate burosumab treatment
4. Have a corrected serum calcium level < 10.8 mg/dL
5. Have an eGFR >25 mL/min/1.73m2 (using CKD-EPI equation)
6. Must be willing in the opinion of the investigators, to comply with study procedures and schedule
7. Provide written informed consent by the subject or a Legal Authorized Representative (LAR) after the study has been explained and prior to any research related procedures begin
8. Must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study.
9. Must be willing to use a highly effective method of contraception for the duration of the study and for at least 12 weeks after the last dose of the study drug. Highly effective methods of contraception include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (e.g., oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (e.g., oral, injectable, implantable), intrauterine device (IUD) or intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, or sexual abstinence (i.e., refraining from heterosexual intercourse during the entire period of risk associated with the study treatments, when this is in line with the preferred and usual lifestyle of the subject)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Concomitant use of active vitamin D (i.e. calcitriol) and/or exogenous phosphate supplementation during burosumab therapy. Subjects will be allowed over the counter Vitamin D should levels drop below <20 ng/ml
2. Blood phosphorus level within or above the normal range while not taking phosphate or active Vitamin D.
3. Severe renal impairment or end-stage renal disease, defined as an eGFR of less than 25 ml/min/1.73m2
4. The use or enrollment in studies using other investigational therapies including other monoclonal antibodies
5. Subject or Legally Authorized Representative not willing or not able to give written informed consent
6. In the investigator's opinion, the subject may not be able to meet all the requirements for study participation
7. History of hypersensitivity to burosumab excipients that in the opinion of the investigator, places the subject at an increased risk of adverse effects
8. Subject has a condition that in the opinion of the investigator could present a concern for subject safety or data interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Serum Phosphorus change | 52 weeks
  Change from baseline over 52 weeks in serum phosphorus with burosumab treatment.

SECONDARY OUTCOMES:
Changes in 1,25(OH)2-Vitamin D | 52 weeks
  Changes from baseline over 52 weeks in 1,25(OH)2-Vitamin D
Changes in tubular reabsorption of phosphate (TRP) | 52 weeks
  Changes from baseline over 52 weeks in tubular reabsorption of phosphate (TRP)
Changes in TmP/GFR (the ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate | 52 weeks
  Changes from baseline over 52 weeks in TmP/GFR (the ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate
Biomechanical Marker | 52 weeks
  Effect of burosumab over 52 weeks on biochemical marker of bone turnover that reflects osteomalacia severity: alkaline phosphatase (ALP).
6-minute walk test | 52 weeks
  Change in walking capacity over 52 weeks as assessed by 6-Minute Walk Test (6MWT)
Sit-to-Stand test (STST) | 2 weeks
  Change in proximal muscle function over 52 weeks as assessed by the Sit-to-Stand test (STST)
Brief Pain Inventory (BPI) | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by Brief Pain Inventory (BPI)
Brief Fatigue Inventory (BFI) | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by Brief Fatigue Inventory (BFI)
SF36 item short health survey (SF-36) | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by SF36 item short health survey (SF-36)
PROMIS Pain Intensity | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by PROMIS Pain Intensity instrument. Pain is rated on a scale of 0-10 where 0 represents no pain and 10 represents the worst possible pain.
PROMIS Pain Interference | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by PROMIS Pain Interference instrument. Responses are aggregated and converted to a T-score from 0-100 where 50 is the mean and every 10 is one standard deviation from the mean.
PROMIS Physical Function with Mobility Aid | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by PROMIS Physical Function with Mobility Aid instrument. Responses are aggregated and converted to a T-score from 0-100 where 50 is the mean and every 10 is one standard deviation from the mean.
PROMIS Fatigue | 52 weeks
  Change in Patient/parent-Reported Outcomes over 52 weeks as assessed by PROMIS Fatigue instrument. Responses are aggregated and converted to a T-score from 0-100 where 50 is the mean and every 10 is one standard deviation from the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tosi, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States